CLINICAL TRIAL: NCT02604472
Title: Stage-specified Concurrent Chemoradiotherapy With or Without Induction Chemotherapy for Locoregionally-advanced Nasopharyngeal Carcinoma - A Retrospective, Population-based Study
Brief Title: Retrospective Investigation of the Impacts of Prognosis for Nasopharyngeal Carcinoma Patients
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, XIANG YANQUN, associate professor, Sun Yat-sen University
Other Study IDs: 2013046
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Malignant Neoplasm of Other Specified Site of Nasopharynx
Keywords: Nasopharyngeal carcinoma; induction chemotherapy; concurrent chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CCRT group: Locoregionally advanced nasopharyngeal carcinoma patients received concurrent chemoradiotherapy
  Interventions: Other: CCRT
- IC+CCRT group: Locoregionally advanced nasopharyngeal carcinoma patients received induction chemotherapy and concurrent chemoradiotherapy
  Interventions: Other: IC+CCRT

INTERVENTIONS:
Other: CCRT — Locoregionally advanced nasopharyngeal carcinoma patients received platinum-based/non-platinum based concurrent chemoradiotherapy.
  Groups: CCRT group
Other: IC+CCRT — Locoregionally advanced nasopharyngeal carcinoma patients received induction chemotherapy and platinum-based/non-platinum based concurrent chemoradiotherapy.
  Groups: IC+CCRT group

SUMMARY:
To investigate whether the additional induction chemotherapy (IC) to concurrent chemoradiotherapy (CCRT) was able to improve overall survival (OS) and disease-free survival (DFS), and to clarify if stage-specified chemoradiotherapy regimens benefit the most for locoregionally advanced NPC.

DETAILED DESCRIPTION:
Data of patients firstly diagnosed NPC from Jan 1st, 1998 to Jun 1st, 2013 were downloaded from Department of Medical Information, Sun Yat-Sen University Cancer Center. Patients were excluded if they had stage I or II disease, no complete medical records, received treatment previously, or without concurrent chemoradiotherapy. Follow-up data is updated on October 1st, 2015.The propensity score-matching (PSM) method was adopted to balance observed covariates between both groups. Propensity scores reflect the conditional probability that is intended to be uniform between patients received CCRT and IC+CCRT based on their baseline characteristics. Matching was performed based on nearest-neighbor matching, and comparing between CCRT and IC+CCRT patients were matched within their respective risk groups.

ELIGIBILITY:
Inclusion Criteria:

1. firstly diagnosed NPC in SYSUCC from Jan 1st, 1998 to Jun 1st, 2013;
2. with complete medical records;
3. received radical RT.

Exclusion Criteria:

1. distant metastasis patients at first diagnosis,
2. recurrent patients,
3. not finishing radiotherapy, missing medical data, death during RT, stage I or II disease,received treatment previously, or without concurrent chemoradiotherapy were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: firstly diagnosed NPC in SYSUCC from Jan 1st, 1998 to Jun 1st, 2013
Sampling Method: Probability Sample
Enrollment: 12206 (Actual)
Dates: Start 1998-01; Primary Completion 2013-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 10 years

SECONDARY OUTCOMES:
disease-free survival | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Guo, MD, PhD, Study Chair — Sun Yat-sen University

REFERENCES:
- [Derived] Xia WX, Liang H, Lv X, Wang L, Ye YF, Ke LR, Xu LH, Guo X, Xiang YQ. Stage-specific concurrent chemoradiotherapy with or without induction chemotherapy for locoregionally advanced nasopharyngeal carcinoma: a retrospective, population-based study. Cancer Manag Res. 2019 Nov 20;11:9813-9827. doi: 10.2147/CMAR.S179139. eCollection 2019. PMID 31819619